CLINICAL TRIAL: NCT04986397
Title: Cold Therapy For Pain Control Among Pediatric Appendectomy Patients: A Randomized Controlled Trial
Brief Title: Cold Therapy for Pediatric Appendectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Heung Bae Kim, Professor of Surgery, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00038266
Record Dates: First submitted 2021-06-15; First posted 2021-08-02 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Cryotherapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cold Therapy & Standard Post Operative Analgesia (Experimental): Patients in the cryotherapy group will have the ice water in their cryotherapy device maintained continuously for 2 days from initial application as this is the reported time of average patient disability and children typically return to school by post-operative day 3. The device will not be placed directly on the skin to minimize tissue damage. An additional protective barrier pad included with the cold therapy device will provide a barrier between the skin and the cooling device. This allows for continuous cooling at a higher target skin temperature. Aside from the cryotherapy, all surgical treatment will be standard of care.
  Interventions: Device: Cold Therapy; Other: Standard of Care
- Standard Post Operative Analgesia (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Cold Therapy — A Breg Polar Care Cube with WrapOn Polar Pad, Back will be filled with ice chips and water per manufacturer instructions and applied to the abdomen.
  Other Names: Breg Polar Care Cube; Cryotherapy
  Arms: Cold Therapy & Standard Post Operative Analgesia
Other: Standard of Care — Standard post-operative analgesia without the use of cryotherapy.

SUMMARY:
This is a randomized control trial to evaluate the efficacy of an FDA approved cold therapy device vs. usual care among children undergoing appendectomy at a large children's hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age of 7 years of older
* Diagnosis of appendicitis and scheduled appendectomy

Exclusion Criteria:

* Neurologic and Decision Impairment
* Chronic opioid dependency
* Planned ICU admission post-operatively
* Reoperation during hospital stay
* Ward of the state
* Non-english and non-spanish speakers

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Intensity Scale | Post operative days 1-3
  The primary outcome variable in this trial is pain score as reported on the Numeric Pain Intensity Scale. These scores will be self-reported (Numerical Pain Intensity Scale, 0-10 visual analog scale with 0 representing no pain and 10 representing the worst pain imaginable) assessed and documented once daily.

SECONDARY OUTCOMES:
Mean Morphine Metabolic Equivalents (MME) | Limited to duration of hospital stay, up to 1 month
  Mean amount of morphine administered throughout the duration of the hospital stay.
Length of Hospital Stay | Duration of stay in hospital post-operatively, up to 1 month
  Length of time stayed in the hospital before being discharged
Time to Return of Tolerating Solid Food | Duration of time until beginning to tolerate solid food, up to 1 month
  Time in days it takes to tolerate solid foods.

OTHER OUTCOMES:
Brief Pain Inventory Short Form | Post operative days 1-3
  Pain diagram to indicate location of pain and 7 Likert-scale questions assessing pain severity and interference with feeling and function, scores ranging from 0 = No pain to 10 = pain as bad as you can imagine assessed just before hospital discharge and once daily.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rentea RM, Peter SDS, Snyder CL. Pediatric appendicitis: state of the art review. Pediatr Surg Int. 2017 Mar;33(3):269-283. doi: 10.1007/s00383-016-3990-2. Epub 2016 Oct 14. PMID 27743024
- [Background] Cairo SB, Calabro KA, Bowdish E, Reilly C, Watt S, Rothstein DH. Variation in postoperative narcotic prescribing after pediatric appendectomy. J Pediatr Surg. 2019 Sep;54(9):1866-1871. doi: 10.1016/j.jpedsurg.2018.11.015. Epub 2019 Feb 7. PMID 30819545
- [Background] Harbaugh CM, Gadepalli SK. Pediatric postoperative opioid prescribing and the opioid crisis. Curr Opin Pediatr. 2019 Jun;31(3):378-385. doi: 10.1097/MOP.0000000000000768. PMID 31090580
- [Background] Watkins AA, Johnson TV, Shrewsberry AB, Nourparvar P, Madni T, Watkins CJ, Feingold PL, Kooby DA, Maithel SK, Staley CA, Master VA. Ice packs reduce postoperative midline incision pain and narcotic use: a randomized controlled trial. J Am Coll Surg. 2014 Sep;219(3):511-7. doi: 10.1016/j.jamcollsurg.2014.03.057. Epub 2014 May 23. PMID 25081937
- [Background] Chumkam A, Pongrojpaw D, Chanthasenanont A, Pattaraarchachai J, Bhamarapravatana K, Suwannarurk K. Cryotherapy Reduced Postoperative Pain in Gynecologic Surgery: A Randomized Controlled Trial. Pain Res Treat. 2019 Mar 4;2019:2405159. doi: 10.1155/2019/2405159. eCollection 2019. PMID 30949366